CLINICAL TRIAL: NCT05005533
Title: The Effect of Respiratory Muscle Strength and Functional Capacity on Posture and Balance in Individuals With Different Phenotypes of Chronic Obstructive Pulmonary Disease
Brief Title: The Effect of Respiratory Muscle Strength and Functional Capacity on Posture and Balance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ceyhun Topcuoğlu, Principal Investigator, Abant Izzet Baysal University
Other Study IDs: AIBU-FTR-CT-05
Record Dates: First submitted 2021-08-07; First posted 2021-08-13 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Respiratory Muscle Strength; Posture; Balance; Functional Capacity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mild and Moderate Severe Group: Individuals with Chronic Obstructive Pulmonary Disease with a Forced Expiratory Volume greater than 50% of the expected value
  Interventions: Other: Observational
- Severe and Very Severe Group: Individuals with Chronic Obstructive Pulmonary Disease whose Forced Expiratory Volume is less than 50% of the expected value
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Chronic Obstructive Pulmonary Disease Severity of Individuals by Chronic Obstructive Pulmonary Disease Assessment Test, shortness of breath Modified Medical Research Council scale, cough related quality of life Leicester Cough Questionnaire, respiratory muscle strength with Maximum Inspiratory and Expiratory Pressure, Posture with Spinal Mouse device, pain with Visual Analog Scale, severity of fatigue Fatigue Physical performance of the lower extremities will be evaluated with the Short Physical Performance Test, functional mobility will be evaluated with the Time Up and Go Test, and balance will be evaluated with the Biodex Balance System

SUMMARY:
As a result of the study, inspiratory muscle strength, posture and physical performance evaluations of individuals with Chronic Obstructive Pulmonary Disease will be made, suggestions will be made to help individual postural smoothness and improve physical performance.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease is a multifaceted disease that results from the interaction between genetic susceptibility and exposure to environmental stimuli. Due to the slow progression and chronic nature of the disease, it creates a growing disease burden on the individual. Considering the data of the Turkish Statistical Institute, the third most common cause of death in Turkey in 2010, 2011 and 2012 was respiratory system diseases. 61.5% of respiratory system deaths in 2012 were due to Chronic Obstructive Pulmonary Disease. Due to the progressive airway obstruction that occurs in Chronic Obstructive Pulmonary Disease, the level of inspiratory muscle strength is restricted and there is an increasing deterioration in the level of functional performance. However, with increasing age, postural problems can be observed in individuals with Chronic Obstructive Pulmonary Disease. Postural problems such as rounded shoulders, increase in thoracic kyphosis and muscle shortness can be observed especially in patients who start to use the auxiliary respiratory muscles continuously due to inspiratory muscle strength. There are few articles investigating the changes in posture, physical performance and inspiratory muscles with the addition of a chronic disease such as Chronic Obstructive Pulmonary Disease to the normal aging process. For this reason, a study titled "The effect of respiratory muscle strength and functional capacity on posture and balance in individuals with Chronic Obstructive Pulmonary Disease with Different Phenotypes" was planned.

As a result of the study, inspiratory muscle strength, posture and physical performance evaluations of individuals with Chronic Obstructive Pulmonary Disease will be made, and suggestions will be made to help individual postural smoothness and improve physical performance.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Chronic Obstructive Pulmonary Disease according to the Global Initiative for Chronic Obstructive Lung Disease criteria
* Not having vision, hearing and speech problems
* Volunteering to participate in the research

Exclusion Criteria:

* Have had major surgery in the past few months
* History of recurrent significant clinical infection
* Having cognitive problems
* Unstable angina, previous myocardial infarction (MI),
* Severe congestive heart failure resistant to medical treatment,
* Having uncontrolled hypertension,
* Get cancer
* Having neurological or musculoskeletal diseases with functional limitations
* Having suffered an injury, such as a sprain, sprain or fracture of the lower extremity in the last 6 months, unable to perform independent ambulation

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic obstructive pulmonary disease is a common, preventable and treatable disease characterized by persistent respiratory symptoms and airway limitation due to airway and/or alveolar abnormality resulting from exposure to harmful gases or particles and many factors that cause abnormal lung development.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
Maximal Inspiratory Pressure | 5 minutes
  Respiratory muscle strength will be assessed by maximal inspiratory pressure. Values in the normal range indicate normal respiratory muscle strength, low values indicate decreased respiratory muscle strength.

SECONDARY OUTCOMES:
Posture Assessment | 5 minutes
  Posture assessment of individuals will be done with the Spinal Mouse device. Individuals will be asked to distribute their weight equally on both lower extremities as much as possible and to stand symmetrically. The angular deviation between each SPINE will be calculated as an angle. While the high angle of deviation indicates that the posture is bad; A low angle of deviation indicates a good posture
Biodex Balance System | 5 minutes
  Balance assessment will be evaluated with the Biodex Balance System. A high values indicates poor balance, and a low values indicates good balance.
Time Up and Go Test | 2 minutes
  Time Up and Go Test is a balance test that is frequently used to evaluate the functional mobility of individuals. High times indicate impaired functional mobility; low times indicate good functional mobility.
Short Physical Performance Test | 5 minutes
  The physical performance of the lower extremities of the individuals will be evaluated with the Short Physical Performance Test. High values indicate deterioration of physical performance; low values indicate good physical performance.
Chronic Obstructive Pulmonary Disease Assessment Test | 2 minutes
  Chronic Obstructive Pulmonary Disease symptoms are assessed with the Chronic Obstructive Pulmonary Disease Evaluation Test. High values indicate poor health; low values indicate good health
Modified Medical Research Council Scale | 2 minutes
  The breath assessment test will be evaluated with the Modified Medical Research Council Scale. High values indicate high dyspnea; low values indicate low dyspnea.
Leicester Cough Questionnaire | 2 minutes
  The cough related quality of life questionnaire will be assessed by the Leicester Cough Questionnaire. Low values indicate poor quality of life associated with cough; high values indicate good quality of life associated with cough
Visual Analog Scale | 2 minutes
  Pain intensity will be evaluated with a visual analog scale. While high values indicate increased pain intensity; low values indicate low pain intensity
Fatigue Severity Scale | 2 minutes
  Fatigue will be evaluated with the Fatigue Severity Scale. High values indicate increased fatigue severity; lower values indicate lower fatigue severity

CONTACTS AND LOCATIONS:
Locations (1):
- Bolu Abant İzzet Baysal University Department of Physiotherapy and Rehabilitation, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No